CLINICAL TRIAL: NCT01620866
Title: A Controlled, Single-blind Pilot Study of EMDR in Bipolar, Subsyndromal Patients With Trauma
Brief Title: A Eye Movement Desensitization Reprocessing (EMDR) Study in Bipolar Traumatized Patients
Acronym: BET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FIDMAG Germanes Hospitalàries (Other)
Responsible Party: Principal Investigator, Benedikt Amann, Senior researcher, FIDMAG Germanes Hospitalàries
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BET-study
Record Dates: First submitted 2012-06-11; First posted 2012-06-15 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Bipolar Disorder; PTSD
Keywords: EMDR; bipolar disorder; trauma; subsyndromal symptoms; PTSD
MeSH Terms: conditions — Bipolar Disorder; Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMDR (Experimental)
  Interventions: Other: Eye Movement Desensitization Reprocessing (EMDR)
- TAU (No Intervention): Treatment as usual (TAU)

INTERVENTIONS:
Other: Eye Movement Desensitization Reprocessing (EMDR) — EMDR is an effective treatment in PTSD but has never been tested in bipolar traumatized patients.
  Arms: EMDR

SUMMARY:
The purpose of this pilot study is whether Eye Movement Desensitization Reprocessing (EMDR), an approved psychotherapy in posttraumatic stress disorder, improves mood, functioning, quality of life, cognition and BDNF levels in subsyndromal bipolar patients with trauma.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I or II disorder following DSM-IV criteria
* Instable, subsyndromal course defined as at evaluation baseline (HAMD > 8 < 15 and/or YMRS > 7 < 14)
* Good adherence to pharmacological treatment
* Major or minor traumatic life-events
* EMDR therapists > 3 years experience
* Able to sign informed consent

Exclusion Criteria:

* Major affective episode in last 3 months
* Active drug abuse/dependency
* Neurological disease
* Suicidal thoughts/ideation
* Prior treatment EMDR
* DES > 25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is a statistically significant reduction in the YMRS and/or HDRS in the EMDR group compared with the TAU group. | 3 months and 6 months
  Patients with subsydromal symptoms, objectified by the YMRS and HDRS, are included in the study. After randomization to EMDR or TAU, group differences in changes in the YMRS and HRDS are measured at visit after intervention (3 months) and at follow-up (6 months). The hypothesize is that the EMDR group will statistically improve in both affective scales when compared to the TAU group.

SECONDARY OUTCOMES:
The EMDR group improves statistically significant in trauma load when compared to TAU. | 3 months and 6 months
  Secondary outcome measure includes changes in trauma scales (IES, CAPS)from baseline to 3 months and 6 months.
The EMDR group improves statistically significant in cognitive tests when compared to TAU. | 3 months and 6 months
  Subjects underwent a neuropsychologcial battery to test various cognitive domains.
The EMDR group improves statistically significant in functioning when compared to TAU. | 3 months and 6 months
  All subjects were evaluated with respect to their functioning using the FAST, a validated scale of functioning in bipolar disorder.
The EMDR group improves statistically significant in quality of life when compared to TAU. | 3 months and 6 months
  Possible changes of Quality of life were tested in all subjects as well, using the SF-36.
Plasma levels of BDNF was statistically higher in the EMDR group after intervention when compared to TAU. | 3 months and 6 months
  Levels of BDNF are lower in bipolar patients, and even lower when traumatized, when compared to the general population. We aimed to find higher levels of BDNF in the EMDR group.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt L Amann, MD, Principal Investigator — FIDMAG Germanes Hospitalàries
Locations (1):
- FIDMAG, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Kauer-Sant'Anna M, Tramontina J, Andreazza AC, Cereser K, da Costa S, Santin A, Yatham LN, Kapczinski F. Traumatic life events in bipolar disorder: impact on BDNF levels and psychopathology. Bipolar Disord. 2007 Jun;9 Suppl 1:128-35. doi: 10.1111/j.1399-5618.2007.00478.x. PMID 17543031
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720